CLINICAL TRIAL: NCT07368439
Title: Effects of Feedback-Based Balance Training on Balance and Gait Performance in Cancer Patients With Chemotherapy-Induced Peripheral Neuropathy (CIPN): A Randomized Controlled Trial
Brief Title: Effect of Feedback-Based Balance Training on Balance and Gait in Cancer Patients With Chemotherapy-Induced Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Amna Zia, Physiotherapist/ Lecturer, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 66/RC/KEMU
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy (CIPN)
Keywords: Chemotherapy-Induced Peripheral Neuropathy; Balance Training; Feedback-Based Training; Gait Training; Physiotherapy; Cancer Rehabilitation; Fall Prevention; Postural Control

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to either an experimental group receiving feedback-based balance training in addition to conventional physiotherapy or a control group receiving conventional physiotherapy alone.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to group allocation by providing both groups with supervised physiotherapy sessions of similar duration and structure, without disclosure of group-specific intervention details. Outcome assessors will be blinded to treatment allocation. Due to the nature of the intervention, care providers delivering the physiotherapy cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback-Based Balance Training Plus Conventional Physiotherapy (Experimental): Participants in this arm will receive conventional physiotherapy combined with feedback-based balance and gait training. Conventional physiotherapy will include strengthening, flexibility, and general balance exercises. Feedback-based balance training will consist of task-oriented balance and gait activities incorporating visual and verbal feedback, mirror-based exercises, and functional gait tasks designed to challenge postural control and coordination. Sessions will be supervised, last approximately 30 minutes, and will be conducted twice per week for four weeks.
  Interventions: Other: Feedback-Based Balance and Gait Training
- Conventional Physiotherapy (Active Comparator): Participants in this arm will receive conventional physiotherapy focused on strengthening, flexibility, and general balance exercises commonly used in the rehabilitation of patients with peripheral neuropathy. Sessions will be supervised, last approximately 30 minutes, and will be conducted twice per week for four weeks.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Feedback-Based Balance and Gait Training — Feedback-based balance and gait training will include structured, task-oriented balance and walking activities designed to challenge postural control and coordination. The intervention will incorporate visual and verbal feedback provided by the therapist, mirror-based exercises, and functional gait tasks such as obstacle negotiation and controlled walking activities. Training will be supervised and delivered in sessions lasting approximately 30 minutes, twice per week for four weeks. This intervention will be provided in addition to conventional physiotherapy.
  Arms: Feedback-Based Balance Training Plus Conventional Physiotherapy
Other: Conventional Physiotherapy — Conventional physiotherapy will include standard rehabilitation exercises commonly used for patients with peripheral neuropathy, such as strengthening exercises, flexibility exercises, and general balance training. Sessions will be supervised by a physiotherapist and delivered for approximately 30 minutes per session, twice per week for four weeks.
  Arms: Conventional Physiotherapy

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common complication of cancer treatment that can cause numbness, tingling, pain, balance problems, and difficulty walking. These symptoms may increase the risk of falls and reduce independence and quality of life in cancer survivors.

The purpose of this study is to determine whether adding feedback-based balance training to conventional physiotherapy improves balance and walking ability in cancer patients with CIPN. Participants will be randomly assigned to one of two groups. One group will receive conventional physiotherapy along with feedback-based balance and gait training, while the other group will receive conventional physiotherapy alone.

The intervention will be provided twice per week for four weeks. Balance, gait performance, neuropathy symptoms, and fear of falling will be assessed before and after the intervention using standardized clinical outcome measures. The findings of this study may help identify effective rehabilitation strategies to improve balance and mobility in cancer patients affected by chemotherapy-induced peripheral neuropathy.

DETAILED DESCRIPTION:
This study is a single-blind, parallel-group randomized controlled trial designed to evaluate the effects of feedback-based balance training on balance and gait performance in cancer patients with chemotherapy-induced peripheral neuropathy (CIPN).

Eligible participants will be adults aged 30 to 60 years with a diagnosis of breast, rectal, or stomach cancer who have developed peripheral neuropathy following neurotoxic chemotherapy. Participants must be able to walk at least six meters independently and demonstrate clinically relevant neuropathy symptoms as measured by the EORTC CIPN20 questionnaire. Individuals with other causes of peripheral neuropathy, significant neurological disorders, severe visual impairment, or musculoskeletal conditions affecting balance will be excluded.

A total of 70 participants will be recruited and randomly allocated into two groups in a 1:1 ratio. The experimental group will receive conventional physiotherapy combined with feedback-based balance and gait training, while the control group will receive conventional physiotherapy alone. Randomization will be performed using a simple random allocation method. Outcome assessors will be blinded to group allocation.

The intervention will be delivered twice weekly for four weeks, with each session lasting approximately 30 minutes. Feedback-based balance training will include task-oriented balance and gait activities incorporating visual and verbal feedback, mirror-based exercises, and functional gait tasks designed to challenge postural control and coordination. Conventional physiotherapy will include strengthening, flexibility, and general balance exercises.

Outcome measures will be assessed at baseline and immediately after completion of the four-week intervention. Primary outcomes include balance performance measured using the Berg Balance Scale and gait performance measured by walking speed. Secondary outcomes include neuropathy-related symptoms assessed using the EORTC CIPN20 questionnaire and fear of falling assessed using the Falls Efficacy Scale-International (FES-I).

This study aims to provide evidence on the effectiveness of feedback-based balance training as an adjunct to conventional physiotherapy for improving balance, gait, and functional confidence in cancer patients with chemotherapy-induced peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 30 to 60 years

Diagnosed with breast, rectal, or stomach cancer

History of treatment with neurotoxic chemotherapy

Presence of chemotherapy-induced peripheral neuropathy as indicated by an EORTC CIPN20 total score of 24 or higher

Ability to walk independently for at least 6 meters, with or without an assistive device

Medically stable and able to participate in physiotherapy

Exclusion Criteria:

* Peripheral neuropathy due to causes other than chemotherapy (e.g., diabetes mellitus)

History of neurological disorders affecting balance or gait (e.g., stroke, Parkinson's disease)

Severe musculoskeletal conditions affecting balance or lower limb function

Active foot ulcers, infections, or soft tissue injuries

Severe visual impairment affecting balance

Any medical condition that, in the investigator's judgment, would interfere with safe participation

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-03-29 (Estimated); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
Balance Performance | Baseline and immediately after completion of the 4-week intervention
  Balance performance will be evaluated using the Berg Balance Scale (BBS), a 14-item standardized clinical assessment with total scores ranging from 0 to 56, where higher scores indicate better balance.

SECONDARY OUTCOMES:
Gait Performance | Baseline and immediately after completion of the 4-week intervention
  Gait performance will be assessed by measuring walking speed over a standardized 6-meter walking distance. Walking speed will be calculated in meters per second, with higher values indicating better gait performance.
Chemotherapy-Induced Peripheral Neuropathy Symptoms | Baseline and immediately after completion of the 4-week intervention
  Severity of chemotherapy-induced peripheral neuropathy symptoms will be assessed using the European Organisation for Research and Treatment of Cancer Chemotherapy-Induced Peripheral Neuropathy questionnaire (EORTC CIPN20). Higher scores indicate greater severity of neuropathy-related symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Amna Zia, PhD. Scholar, Principal Investigator — King Edward Medical University, Lahore; Muhammad Saad Khalid, Principal Investigator — King Edward Medical University, Lahore; Rizwan Haider, PhD. Scholar, Study Director — King Edward Medical University, Lahore
Locations (1):
- King Edward Medical University, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly due to the single-center nature of the study, institutional data protection policies, and the absence of participant consent for public data sharing. De-identified, aggregated results will be reported in publications and presentations.

REFERENCES:
- [Background] Yardley L, Beyer N, Hauer K, Kempen G, Piot-Ziegler C, Todd C. Development and initial validation of the Falls Efficacy Scale-International (FES-I). Age Ageing. 2005 Nov;34(6):614-9. doi: 10.1093/ageing/afi196. PMID 16267188
- [Background] Staff NP, Grisold A, Grisold W, Windebank AJ. Chemotherapy-induced peripheral neuropathy: A current review. Ann Neurol. 2017 Jun;81(6):772-781. doi: 10.1002/ana.24951. Epub 2017 Jun 5. PMID 28486769
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Maki B. Measuring balance in the elderly: validation of an instrument. Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S7-11. PMID 1468055